## STUDY PROTOCOL

| The Effect | of Balint-Based | Group | Intervention | on Burnout | and | Communication | Skills | in |
|---|---|---|---|---|---|---|---|---|
| Nurses | | | | | | | | |

Sponsor / Responsible Party:

Reyhan Doğan, PhD, RN

Bilecik Şeyh Edebali University, Faculty of Health Sciences

Study Type:

Two-arm Parallel Randomized Controlled Trial

NCT Number: XXXX

Document Type: Study Protocol With Statistical Analysis Plan And Informed Consent Form

Document Date: 19 September 2024

Version: Version 1.0

## INFORMED CONSENT FORM

You have been invited to participate in a study titled "The Effect of Balint Approach Group Intervention on Burnout and Communication Skills in Nurses." Participation in the study is voluntary. This form has been prepared to obtain your consent to collect certain information about you for the purposes of this research. If you agree to participate in the study, you will not incur any financial obligations, and you will not be paid. You have the right to withdraw from the study at any time. If you consent to the use of your information for scientific purposes, provided that your identity remains confidential, you will be asked to sign this form. The information obtained from this study will be used for research purposes, and your personal information will be kept confidential. To achieve the purpose of the study, you are expected to provide complete and accurate answers to the questions asked. If you require further information beyond what is provided in this research, you may contact the responsible researcher, Dr. Reyhan DOĞAN, now or send an email to reyhan.dogan@yiu.edu.tr.

## (Participant's Declaration)

Dr. Reyhan DOĞAN, an Assistant Professor at Yüksek İhtisas University, informed me that a medical research study would be conducted and shared the above information with me. I read the relevant text. Following this information, I was invited to participate in this research as a "participant."

I have not encountered any coercive behavior regarding my participation in the research. I also know that if I refuse to participate, this will not harm my patient-nurse relationship in any way. I can withdraw from the research at any time during the project without giving any reason (however, I am aware that it would be appropriate to inform the researchers in advance that I will withdraw from the research so as not to put them in a difficult position). I am not assuming any financial responsibility for the expenses incurred for the research. I will not be paid.

I fully understand all the explanations given to me. I agree to participate in the research in question with my own consent, without any pressure or coercion, on a voluntary basis, under these conditions. A copy of this signed form will be given to me.

| Participant's Name and Surname: | Principal investigator |
|---------------------------------|------------------------|
| Address: | Address: |
| Phone: | Tel: |
| Signature: | Signature: |
| Date: | Date |